CLINICAL TRIAL: NCT03278483
Title: Efficacy, Security, Adherence, Tolerability and Cost Effectiveness of Latent TB Treatment in Patients With TB/DM2
Brief Title: Efficacy, Security, Adherence, Tolerability and Cost Effectiveness of Latent TB Treatment in Patients With TB/DM2 (TBL)
Acronym: TBL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Nacional de Salud Publica, Mexico (Other)
Collaborators: Instituto Nacional de Enfermedades Respiratorias (Other Government); Instituto Nacional de Ciencias Medicas y Nutrición (Unknown)
Responsible Party: Principal Investigator, Ma. de Lourdes Garcia Garcia, Director of prevention of infectious diseases, Instituto Nacional de Salud Publica, Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1341
Record Dates: First submitted 2017-08-07; First posted 2017-09-11 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Diabetes Mellitus; Tuberculin (Skin Test) Positive
Keywords: Latent tuberculosis, ,; isoniazid, rifampin,; rifampin,; adverse,; diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus; Latent Tuberculosis | interventions — Isoniazid; Tablets; Isonicotinic Acids; Rifampin

STUDY DESIGN:
Intervention Model Description: * Arm Isoniacid Diabetic patients with a positive TST of >10mm, who wil be randomly assigned to receive treatment with isoniazid tablets 300mg daily plus pyridoxine 50mg daily
  * Arm B Diabetic patients with a positive TST of >10mm, who wil be randomly assigned to receive treatment with rifampin capsules 600mg daily
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Isoniazid (Active Comparator): Diabetic patients with a positive TST of >10mm, will be randomly assigned to receive treatment with isoniazid 300mg Oral Tablet daily plus pyridoxine 50mg daily for six months
  Interventions: Drug: Isoniazid 300 mg Oral Tablet
- Rifampin (Active Comparator): Diabetic patients with a positive TST of >10mm, who wil be randomly assigned to receive treatment with rifampin 600mg Oral Tablets daily for three months
  Interventions: Drug: Rifampin 600 mg Oral Tablet

INTERVENTIONS:
Drug: Isoniazid 300 mg Oral Tablet — Isoniazid tablets 300mg daily plus pyridoxine 50mg daily
  Other Names: Isonicotinic acid
  Arms: Isoniazid
Drug: Rifampin 600 mg Oral Tablet — Rifampin capsules 600mg daily
  Other Names: Rifadin
  Arms: Rifampin

SUMMARY:
Researchers will evaluate the efficacy, toxicity, adherence and cost effectiveness of treatment with isoniazid or rifampicin in patients with diabetes mellitus type two (DM2) and latent TB (LTB).

This is a collaborative study with participation from three national institutes (Instituto Nacional de Salud Pública (INSP), Instituto Nacional de Enfermedades Respiratorias (INER) and the Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubiran (INCMNSZ)).

The study will take place in the VII sanitary jurisdiction of Orizaba and the INCMNSZ that has the necessary infrastructure and human resources. Researchers will evaluate 3000 patients with diabetes using a standardized questionnaire and a tuberculin skin test (TST) test. Eligible patients will be invited to participate and from those that agree to participate and sign a written informed consent we will obtain clinical, epidemiological, nutritional and metabolic information. Patients with altered liver function tests will be excluded.

DETAILED DESCRIPTION:
This study is a randomized control trial, with two parallel arms, fixed assignment, fixed sample size and in two study sites. Participants will be assigned 1:1 to receive one of the two treatment regimens: isoniazid for 6 months or rifampicin for 3 months. The assignment will be fixed because the covariates that predict the clinical outcome and the accumulated outcome of participants will not affect treatment assignment. In patients that the Michigan evaluation identifies as having neuropathic changes researchers will perform an electroneurography in order to identify the degree of neuropathy if any. This will be performed in the neurophysiology lab of the INCMNSZ. An independent comity will monitor adverse events.

Sample size It is necessary to include 193 participants, for each arm; this includes a 20% increase to compensate loss during follow up. This will provide a power equal or higher than 80% considering an alpha of 0.05 (.25 at two tails) in order to answer to each one of the following objectives.

Latent tuberculosis treatment with isoniazid is the gold standard and given its efficacy it would not be ethical to propose a placebo group. Researchers hypothesize that treatment with rifampicin will not be inferior in efficacy (measured using the response of biomarkers) and will be equivalent in toxicity to that observed with isoniazid treatment.

Subjects will be asked to attend on the 15th and 30th of the month and then once a month till the end of treatment. In case a patient does not assist, researchers will carry out a home visit.

Clinical, microbiological and metabolic evaluation

Researchers will apply a validated questionnaire that explores sociodemographic, epidemiological and clinical information as well as a questionnaire developed by the researchers that captures information of DM2 long term complications. The Michigan questionnaire will be applied using the NCI-CTC scale in version 3 for neuropathic symptoms as well as an evaluation with a Semmes-Weinstein monofilament of 5.07/10gr in 4 points of the sole of each foot:

* Distal phalange of the 1st toe, base of the 1st metatarsal and base of the 3rd metatarsal
* Base of the 5th metatarsal In a subsample researchers will carry out an electroneurography study in order to measure and document the level of likely damage as an adverse event.

Tuberculin Skin Test (TST) In patients with DM2 researchers will apply TST using the Mantoux technique. Reactivity will be measured with the diameter of the induration at 48 and 72 hours. Patients with a TST>10mm will be randomized to the trail.

Chest X ray All patients with a positive TST will have a chest X ray taken which will be evaluated by a pulmonologist in order to exclude millar TB.

All patients will be tested for hematic cytology, glucose, glycosylated hemoglobin, and creatinine and liver tests. All lab tests will be carried out using standardized methods that are commercially available.

All documentation of clinical evaluations will be included in the patient's medical chart. These will be safeguarded by the main researcher and confidentiality will be protected at all times.

TB tests During follow up respiratory symptoms will be evaluated. Patients with respiratory symptoms of more than 2 weeks will be asked to give 3 sputum samples in order to analyze for acid fast bacilli (AFB) and Mycobacterium tuberculosis (MTB) culture using standardized methods.

All samples will be identified with a code that links the sample with clinical and epidemiological data. Researchers have established a system that prevents unauthorized people from accessing the samples and personal data.

Field work Personnel have been trained in the good clinical practice course which Works very closely with the health centers. Activities are monitored by supervisors that have been trained to insure the coordination of activities and quality control.

Independent comity for monitoring adverse events For this study researchers will integrate an independent comity to monitor adverse events, which will revise all adverse events and will give follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes mellitus (DM2) diagnosed based on the National Official Norm
2. respiratory symptoms
3. Tuberculin Skin Test (TST) >10mm of induration
4. chest X ray without pleural, lung or mediastinal lesions
5. hemoglobin < 8 gm/dl
6. platelets > 60,000 per microliter
7. bilirubin < 2.5 mg/dl
8. Aspartate aminotransferase (AST) , Glutamic oxalacetic transaminases (SGOT) and alkaline phosphatase less than twice the normal value
9. negative pregnancy test
10. negative Human immunodeficiency virus infection test (HIV test)
11. signed written informed consent.

Exclusion Criteria:

1. Attending selected cites
2. Respiratory symptoms defined as cough with or without sputum for more than 2 weeks
3. Evidence or clinical suspicion of active tuberculosis (TB)
4. Current treatment with antituberculous drugs
5. History of having received more than one month's treatment for latent Tuberculosis (LTB) or antituberculous drugs
6. Hypersensitivity or intolerance to isoniazid or rifampicin
7. Active hepatopathy
8. Grade III or higher peripheral neuropathy
9. Chronic alcohol ingestion
10. Contacts of patients with isoniazid or rifampicin drug resistance

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Efficacy of treatment with rifampicin compared to efficacy of treatment with isoniazid | Up to 18 months
  Researchers will measure with ELISA in vitro production of interferon gamma of peripheric mononuclear cels as a response to stimuli by RV0849 and RV1737 antigens. The cut of value is of >100pg/ml.
Toxicity (neuropathy) | Up to 6 months
  Neurological alterations will be assessed using the Michigan questionnaire and in a subsample they will evaluate neuropathy using electroneurography.
Adherence | Up to 6 months
  Counting the number of administered pills, adequate adherence is more than 80% of administered pills.
Toxicity (liver function) | Up to 6 months
  Liver function tests

CONTACTS AND LOCATIONS:
Overall Officials: Jose JS Sifuentes -Osornio, Dr, Principal Investigator — Instituto Nacional de Ciencias Médcias y Nutrición; Martha MT Torres-Rojas, DCs, Principal Investigator — Instituto Nacional de Enfermedades Respiratorias
Locations (1):
- Instituto Nacional de Ciencias Medicas y Nutrición, Mexico City, Mexico

REFERENCES:
- [Result] Torres M, Garcia-Garcia L, Cruz-Hervert P, Guio H, Carranza C, Ferreyra-Reyes L, Canizales S, Molina S, Ferreira-Guerrero E, Tellez N, Montero-Campos R, Delgado-Sanchez G, Mongua-Rodriguez N, Sifuentes-Osornio J, Ponce-de Leon A, Sada E, Young DB, Wilkinson RJ. Effect of isoniazid on antigen-specific interferon-gamma secretion in latent tuberculosis. Eur Respir J. 2015 Feb;45(2):473-82. doi: 10.1183/09031936.00123314. Epub 2014 Oct 30. PMID 25359354